CLINICAL TRIAL: NCT00279877
Title: Cost Effectiveness and Efficacy of Kypho and Vertebro Plasty Trial
Brief Title: Cost Effectiveness and Efficacy of Kyphoplasty and Vertebroplasty Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Cardinal Health (Industry); ArthroCare Corporation (Other); Cook Group Incorporated (Industry)
Responsible Party: Principal Investigator, Avery Evans, MD, MD, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12031
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Osteoporotic Vertebral Compression Fractures
MeSH Terms: interventions — Kyphoplasty

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- vertebroplasty (Active Comparator): vertebroplasty
  Interventions: Procedure: Kyphoplasty
- kyphoplasty (Active Comparator): kyphoplasty
  Interventions: Procedure: Kyphoplasty

INTERVENTIONS:
Procedure: Kyphoplasty — kyphoplasty

SUMMARY:
Randomized trial comparing cost effectiveness and efficacy of kyphoplasty vs vertebroplasty for the treatment of painful, osteoporotic vertebral compression fractures.

ELIGIBILITY:
* > or = 50 years of age
* Compression fracture (T4-L5)within previous 12 mo.
* Pain from compression fracture
* No malignant tumor
* No back surgery

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2005-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Back specific functional status(Roland) | 12 mo
Pain | 12 mo

SECONDARY OUTCOMES:
Health status outcome measure(SF-36) | 12 mo

CONTACTS AND LOCATIONS:
Overall Officials: Avery Evans, M.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Evans AJ, Kip KE, Brinjikji W, Layton KF, Jensen ML, Gaughen JR, Kallmes DF. Randomized controlled trial of vertebroplasty versus kyphoplasty in the treatment of vertebral compression fractures. J Neurointerv Surg. 2016 Jul;8(7):756-63. doi: 10.1136/neurintsurg-2015-011811. Epub 2015 Jun 24. PMID 26109687